CLINICAL TRIAL: NCT00137449
Title: A Phase 2 Efficacy And Safety Study Of SU011248 Administered In A Continuous Daily Regimen In Patients With Advanced Gastrointestinal Stromal Tumor
Brief Title: Study Of SU011248 Administered On A Continuous Daily Dosing Schedule In Patients With Gastrointestinal Stromal Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181047
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Results first posted 2009-09-04 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: SU011248

INTERVENTIONS:
Drug: SU011248 — 37.5 mg once daily on a continuous daily dosing schedule. Study medication continued as long as patient was obtaining clinical benefit, or until significant toxicity, or withdrawal of consent, for up to 1 year on study.

SUMMARY:
To evaluate the antitumor activity of SU011248 in advanced, imatinib mesylate-resistant gastrointestinal stromal tumor (GIST) when administered on a continuous daily dosing schedule

DETAILED DESCRIPTION:
Subjects experiencing clinical benefit after 1 year on study were offered continued treatment with SU011248 on a separate protocol.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven diagnosis of malignant GIST that was not amenable to standard therapy.
* Failed prior treatment with imatinib mesylate, defined either by progression of disease (according to Response Evaluation Criterion in Solid Tumors (RECIST) or World Health Organization (WHO) criteria), or by significant toxicity during treatment with imatinib mesylate that precluded further treatment. Intolerance to prior imatinib mesylate therapy was defined as follows:
* Life-threatening adverse events (ie, Grade 4) at any dose (attempt to dose reduce or rechallenge not required) or Unacceptable toxicity induced by a moderate dose (eg, 400 mg/day), specifically, Grade 2 toxicity that was unacceptable to the patient (such as nausea) that persisted despite standard countermeasures
* Evidence of unidimensionally measurable disease.

Exclusion Criteria:

* Previous treatment on a SU011248 clinical trial.
* Diagnosis of any second malignancy within the last 3 years, except basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma, that had been adequately treated with no evidence of recurrent disease for 12 months.
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease.
* Any of the following within the 12 months prior to starting the study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of grade 2, atrial fibrillation of any grade, or QTc interval >450 msec for males or >470 msec for females.
* Hypertension that could not be controlled by medications (>150/100 mm/Hg despite optimal medical therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Pfizer Investigational Site, Boston, Massachusetts, United States
- France (2):
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Villejuif
- Pfizer Investigational Site, Milan, Italy

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181047&StudyName=Study%20Of%20SU011248%20Administered%20In%20A%20Daily%20Regimen%20In%20Patients%20With%20Gastrointestinal%20Stromal%20Tumor

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Must have failed prior treatment with imatinib mesylate (IM) [defined as progression of disease using Response Evaluation Criteria in Solid Tumors(RECIST) or World Health Organization(WHO) criteria, or significant toxicity during treatment with IM precluding further treatment & Eastern Cooperative Oncology Group(ECOG) performance status of 0-1]
Groups:
- AM Dose Sunitinib Malate; PM Dose Sunitinib Malate: Subjects received sunitinib malate at a starting dose of 37.5 mg/day in repeated 4-week cycles and cycles could be repeated for up to 1 year in the absence of any withdrawal criteria. Subjects were randomized to receive either morning (AM) or afternoon (PM) dose. Doses could be increased to 50 mg daily.
Period: Overall Study
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate
Started | 30 | 30
Completed | 14 | 12
Not Completed | 16 | 18
Not completed — Disease Progression | 8 | 13
Not completed — Death | 4 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 17 | 18 | 35.0
  >=65 years | 13 | 12 | 25.0
Age Continuous [Mean (Standard Deviation); unit: years] | 59.3 (14.5) | 57.0 (14.8) | 58.2 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32.0
  Male | 15 | 13 | 28.0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Benefit Response (CBR) According to RECIST
Description: CBR is defined as a confirmed complete response (CR), confirmed partial response (PR), or stable disease (SD) for at least 24 weeks on study according to RECIST. Confirmed responses are those that persisted on repeat imaging >= 4 wks after initial response. Participants with no on-study radiographic tumor re-evaluation counted as non-responders.
Time Frame: Planned duration on this protocol of up to 1 year
Population: ITT population (all subjects enrolled that received at least 1 dose of study medication) with measurable disease at baseline and correct histological cancer type. CR+PR+(SD for >=24 weeks)
Measure: Number; unit: participants
Groups:
- Total (Equals AM Plus PM Dose) Sunitinib Malate: Subjects received sunitinib malate at a starting dose of 37.5 mg/day in repeated 4-week cycles and cycles could be repeated for up to 1 year in the absence of any withdrawal criteria. Subjects were randomized to receive either morning (AM) or afternoon (PM) dose. Doses could be increased to 50 mg daily.
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate | Total (Equals AM Plus PM Dose) Sunitinib Malate
Number analyzed (Participants) | 30 | 30 | 60
participants | 15 [31.3 to 68.7] | 17 | 32
Statistical Analysis 1: Comparison: AM Dose Sunitinib Malate; Test type: Superiority or Other; F distribution; CBR Rate (percentage) = 50.0, 95% CI [31.3 to 68.7]
Statistical Analysis 2: Comparison: PM Dose Sunitinib Malate; Test type: Superiority or Other; F distribution; CBR Rate (percentage) = 56.7, 95% CI [37.4 to 74.5]
Statistical Analysis 3: Comparison: Total (Equals AM Plus PM Dose) Sunitinib Malate; Null hypothesis that the true CBR <=20% vs the alternative hypothesis that the true clinical benefit rate is at least 35%. The sample size is determined using a single-stage design with an alpha level of 10% & 90% power. If >=17 CR, PR or SD for at least 24 weeks are observed, null hypothesis can be rejected with a 20% target false positive error rate. If <= 16 CR, PR,or SD for at least 24 weeks are observed, null hypothesis can not be rejected with a target false negative error rate of 10%; Test type: Superiority or Other; F distribution; CBR Rate (percentage) = 53.3, 95% CI [40.0 to 66.3]

2. Secondary Outcome: Number of Participants by Best Confirmed Response Category According to RECIST
Description: Best confirmed response (BCR) defined as best response [confirmed CR, confirmed PR, SD, PD(progressive disease), not evaluable (NE)] recorded from start of treatment until disease progression / recurrence. Best response of SD must have met SD criteria at least once after first dose at minimum interval of 6 weeks.
Time Frame: Planned duration on this protocol of up to 1 year
Population: ITT population (all subjects enrolled that received at least 1 dose of study medication) with measurable disease at baseline and correct histological cancer type.
Measure: Number; unit: participants
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate | Total (Equals AM Plus PM Dose) Sunitinib Malate
Number analyzed (Participants) | 30 | 30 | 60
participants
  Complete Response (CR) | 0 | 0 | 0
  Partial Response (PR) | 3 | 5 | 8
  Stable Disease (SD) | 20 | 20 | 40
  Progressive disease (PD) | 2 | 4 | 6
  Not evaluable (NE) | 5 | 1 | 6

3. Secondary Outcome: Number of Participants With Overall Confirmed Objective Disease Response (ORR)
Description: Overall confirmed objective disease response is defined as a confirmed CR, or confirmed PR according to RECIST. Confirmed responses are those that persisted on repeat imaging >= 4 wks after initial response.
Time Frame: Planned duration on this protocol of up to 1 year
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate | Total (Equals AM Plus PM Dose) Sunitinib Malate
Number analyzed (Participants) | 30 | 30 | 60
participants | 3 | 5 | 8
Statistical Analysis 1: Comparison: AM Dose Sunitinib Malate; Test type: Superiority or Other; F distribution; ORR rate (percentage) = 10.0, 95% CI [2.1 to 26.5] — PR or CR responding tumor measurements confirmed by repeat studies performed at > 4 weeks after the criteria for response first met
Statistical Analysis 2: Comparison: PM Dose Sunitinib Malate; Test type: Superiority or Other; F distribution; ORR rate (percentage) = 16.7, 95% CI [5.6 to 34.7] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Total (Equals AM Plus PM Dose) Sunitinib Malate; Test type: Superiority or Other; F distribution; ORR rate (percentage) = 13.3, 95% CI [5.9 to 24.6] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Duration of Stable Disease
Description: Duration of SD is the time from the date of first documentation of stable disease to the date of first documentation of objective tumor progression or death due to any cause that occurred within 28 days after last dose of study medication, whichever occurred first.
Time Frame: Planned duration on this protocol of up to 1 year
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate | Total (Equals AM Plus PM Dose) Sunitinib Malate
Number analyzed (Participants) | 30 | 30 | 60
Participants
  >= 12 weeks | 19 | 14 | 33
  >= 24 weeks | 12 | 12 | 24

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of first dose of study medication to the date of first documentation of objective tumor progression or to death due to any cause that occurred on treatment including within 28 days after the last dose of study medication, whichever occurred first.
Time Frame: Planned duration on this protocol of up to 1 year
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate | Total (Equals AM Plus PM Dose) Sunitinib Malate
Number analyzed (Participants) | 30 | 30 | 60
participants
  Patient was censored | 12 | 10 | 22
  Patient observed to have an event | 18 | 20 | 38
Statistical Analysis 1: Comparison: AM Dose Sunitinib Malate; 95% CI calculated based on the method of Brookmeyer and Crowley. Median reported is progression free survival weeks; Test type: Superiority or Other; Kaplan-Meier method; median = 27.0, 95% CI [22.0 to 73.1]
Statistical Analysis 2: Comparison: PM Dose Sunitinib Malate; 95% CI calculated based on the method of Brookmeyer and Crowley.Median reported is progression free survival weeks; Test type: Superiority or Other; Kaplan-Meier method; median = 35.1, 95% CI [24.4 to 51.6]
Statistical Analysis 3: Comparison: Total (Equals AM Plus PM Dose) Sunitinib Malate; 95% CI calculated based on the method of Brookmeyer and Crowley.Median reported is progression free survival weeks; Test type: Superiority or Other; Kaplan-Meier method; median = 33.6, 95% CI [24.1 to 49.0]

6. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as the time from the date of first dose of study medication to the date of first documentation of objective tumor progression that occurred on treatment including within 28 days after the last dose of study medication.
Time Frame: Planned duration on this protocol of up to 1 year
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate | Total (Equals AM Plus PM Dose) Sunitinib Malate
Number analyzed (Participants) | 30 | 30 | 60
participants
  Patient was censored | 18 | 13 | 31
  Patient observed to have an event | 12 | 17 | 29
Statistical Analysis 1: Comparison: AM Dose Sunitinib Malate; 95% CI calculated based on the method of Brookmeyer and Crowley.Time to progression in weeks reported as median; Test type: Superiority or Other; Kaplan-Meier method; median = 57, 95% CI [24.1 to 73.1]
Statistical Analysis 2: Comparison: PM Dose Sunitinib Malate; 95% CI calculated based on the method of Brookmeyer and Crowley.Time to progression in weeks reported as median; Test type: Superiority or Other; Kaplan-Meier method; median = 42.1, 95% CI [26.1 to 65.9]
Statistical Analysis 3: Comparison: Total (Equals AM Plus PM Dose) Sunitinib Malate; 95% CI calculated based on the method of Brookmeyer and Crowley.Time to progression in weeks reported as median; Test type: Superiority or Other; Kaplan-Meier method; median = 42.1, 95% CI [26.1 to 65.9]

7. Secondary Outcome: Duration of Tumor Response (DR) [Descriptive Statistics]
Description: DR was defined as the time from the date of first documentation of objective tumor response (CR or PR) that was subsequently confirmed to the date of the first documentation of objective tumor progression or to death due to any cause that occurred within 28 days after the last dose of study medication, whichever occurred first.
Time Frame: Planned duration on this protocol of up to 1 year
Population: ITT population (all subjects enrolled that received at least 1 dose of study medication) with measurable disease at baseline and correct histological cancer type. Number of responders (AM=3, PM=5, Total=8)
Measure: Median (Full Range); unit: weeks
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate | Total (Equals AM Plus PM Dose) Sunitinib Malate
Number analyzed (Participants) | 30 | 30 | 60
weeks | 32.7 [32.3 to 35.1] | 40.3 [17.1 to 51.4] | 33.9 [17.1 to 51.4]

8. Secondary Outcome: Overall Survival (OS) and One-year Survival [Descriptive Statistics]
Description: Overall survival is defined as time from the date of first dose of study medication to the date of death due to any cause. One year survival rate defined as the probability that a patient is alive 1 year after the date of first study medication.
Time Frame: Survival status was collected by telephone contact every 2 months for up to 2 years from study entry.
Population: ITT population (all subjects enrolled that received at least 1 dose of study medication).
Measure: Number; unit: participants
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate | Total (Equals AM Plus PM Dose) Sunitinib Malate
Number analyzed (Participants) | 30 | 30 | 60
participants
  Number of subjects alive | 16 | 17 | 33
  Number of subjects dead | 14 | 13 | 27
Statistical Analysis 1: Comparison: AM Dose Sunitinib Malate; Test type: Superiority or Other; Kaplan-Meier method; 1 year survival rate = 60.0, 95% CI [40.5 to 75.0]
Statistical Analysis 2: Comparison: PM Dose Sunitinib Malate; Test type: Superiority or Other; Kaplan-Meier method; 1 year survival rate = 79.7, 95% CI [60.3 to 90.3]
Statistical Analysis 3: Comparison: Total (Equals AM Plus PM Dose) Sunitinib Malate; Test type: Superiority or Other; Kaplan-Meier method; 1 year survival rate = 69.7, 95% CI [56.3 to 79.7]

9. Secondary Outcome: Score of FACIT-Fatigue Scale
Description: FACIT-Fatigue Scale: Overall score from 13-question questionnaire (measures fatigue/asthenia for patients with chronic, life-threatening illnesses). For each question, patient rates condition for the past week on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). Maximum, minimum mean included data available for >=10 subjects.
Time Frame: Baseline, Day 1 & 15 of each treatment cycle
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate | Total (Equals AM Plus PM Dose) Sunitinib Malate
Number analyzed (Participants) | 30 | 30 | 60
score on scale
  Baseline Score | 35.9 (11.13) | 36.3 (13.69) | 36.1 (12.35)
  Maximum Post-Baseline Score | 40.6 (10.38) | 42.8 (8.61) | 41.7 (9.50)
  Minimum Post-Baseline Score | 26.9 (12.39) | 26.0 (13.87) | 26.4 (13.06)

10. Secondary Outcome: Score of EQ-VAS (Euro Quality of Life -Visual Analog Scale)
Description: EQ-VAS score on the self-rated "thermometer," indicating the patient's own assessment of their health status from 0 (worst) to 100 (best) imaginable health state. Change: median score at observation minus median score at baseline. Maximum changes (Increase or Decrease from baseline) included data available for >=10 subjects.
Time Frame: Baseline, Day 1 &15 of each treatment cycle up to 1 year on study
Population: ITT population.
Measure: Median (Full Range); unit: score on scale
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate | Total (Equals AM Plus PM Dose) Sunitinib Malate
Number analyzed (Participants) | 30 | 30 | 60
score on scale
  Maximum Increase | 7.5 [-68.6 to 45.0] | 10.0 [-40.0 to 62.0] | 18.0 [-30.0 to 55.0]
  Maximum Decrease | 0.0 [-80.8 to 50.0] | -10.0 [-30.0 to 67.0] | -7.5 [-80.8 to 62.0]

11. Secondary Outcome: Score of EQ-5D (Euro Quality of Life-5 Dimension) Weighted Health Index
Description: EQ-5D: health status in 5 dimensions (mobility, self-care, pain/discomfort, anxiety/depression, usual activities) with a weighted health Index based on general population values where 0.0 = death and 1.0 = perfect health. Change: median index score at observation minus median index score at baseline (includes data available for >=10 subjects).
Time Frame: Baseline, Day 1 & 15 of each treatment cycle up to 1 year on study
Population: ITT population
Measure: Median (Full Range); unit: score on scale
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate | Total (Equals AM Plus PM Dose) Sunitinib Malate
Number analyzed (Participants) | 30 | 30 | 60
score on scale
  Maximum Increase | 0.1 [-0.2 to 0.7] | 0.0 [-0.6 to 0.8] | 0.1 [-0.4 to 0.8]
  Maximum Decrease | -0.1 [-0.3 to 0.3] | -0.8 [-0.8 to 0.5] | -0.1 [-0.8 to 0.3]

ADVERSE EVENTS:
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 13 | 12
Other Adverse Events (participants affected / at risk) | 30 | 30
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate
Anaemia (Blood and lymphatic system disorders) | 3/30 | 0/30
Vomiting (Gastrointestinal disorders) | 4/30 | 1/30
Diarrhoea (Gastrointestinal disorders) | 3/30 | 0/30
Nausea (Gastrointestinal disorders) | 2/30 | 1/30
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/30 | 1/30
Abdominal pain (Gastrointestinal disorders) | 0/30 | 1/30
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1/30 | 0/30
Constipation (Gastrointestinal disorders) | 0/30 | 1/30
Dental caries (Gastrointestinal disorders) | 0/30 | 1/30
Gastrointestinal perforation (Gastrointestinal disorders) | 1/30 | 0/30
Intestinal obstruction (Gastrointestinal disorders) | 0/30 | 1/30
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0/30 | 1/30
Peritonitis (Gastrointestinal disorders) | 1/30 | 0/30
Pneumatosis intestinalis (Gastrointestinal disorders) | 0/30 | 1/30
Disease progression (General disorders) | 1/30 | 3/30
Asthenia (General disorders) | 3/30 | 0/30
General physical health deterioration (General disorders) | 3/30 | 0/30
Pyrexia (General disorders) | 0/30 | 2/30
Chest pain (General disorders) | 0/30 | 1/30
Chills (General disorders) | 0/30 | 1/30
Death (General disorders) | 1/30 | 0/30
Fatigue (General disorders) | 1/30 | 0/30
Hernia pain (General disorders) | 1/30 | 0/30
Wound infection (Infections and infestations) | 1/30 | 1/30
Catheter related infection (Infections and infestations) | 0/30 | 1/30
Emphysematous cystitis (Infections and infestations) | 0/30 | 1/30
Pyelonephritis (Infections and infestations) | 0/30 | 1/30
Sepsis (Infections and infestations) | 0/30 | 1/30
Septic shock (Infections and infestations) | 1/30 | 0/30
Urinary tract infection (Infections and infestations) | 0/30 | 1/30
Urinary tract infection staphylococcal (Infections and infestations) | 1/30 | 0/30
Blood thyroid stimulating hormone increased (Investigations) | 1/30 | 0/30
Weight decreased (Investigations) | 0/30 | 1/30
Dehydration (Metabolism and nutrition disorders) | 1/30 | 1/30
Anorexia (Metabolism and nutrition disorders) | 1/30 | 0/30
Cachexia (Metabolism and nutrition disorders) | 1/30 | 0/30
Back pain (Musculoskeletal and connective tissue disorders) | 0/30 | 1/30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/30 | 0/30
Cerebrovascular accident (Nervous system disorders) | 0/30 | 1/30
Syncope (Nervous system disorders) | 1/30 | 0/30
Transient ischaemic attack (Nervous system disorders) | 0/30 | 1/30
Confusional state (Psychiatric disorders) | 1/30 | 0/30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate
Anaemia (Blood and lymphatic system disorders) | 15/30 | 14/30
Neutropenia (Blood and lymphatic system disorders) | 9/30 | 9/30
Thrombocytopenia (Blood and lymphatic system disorders) | 7/30 | 6/30
Leukopenia (Blood and lymphatic system disorders) | 4/30 | 2/30
Lymphopenia (Blood and lymphatic system disorders) | 1/30 | 0/30
Macrocytosis (Blood and lymphatic system disorders) | 1/30 | 0/30
Angina pectoris (Cardiac disorders) | 0/30 | 1/30
Palpitations (Cardiac disorders) | 1/30 | 0/30
Ear pain (Ear and labyrinth disorders) | 1/30 | 2/30
Vertigo (Ear and labyrinth disorders) | 2/30 | 1/30
Hypothyroidism (Endocrine disorders) | 4/30 | 4/30
Hyperthyroidism (Endocrine disorders) | 1/30 | 1/30
Eyelash discolouration (Eye disorders) | 1/30 | 3/30
Conjunctival haemorrhage (Eye disorders) | 1/30 | 0/30
Conjunctivitis (Eye disorders) | 1/30 | 0/30
Diplopia (Eye disorders) | 1/30 | 0/30
Eye pruritus (Eye disorders) | 0/30 | 1/30
Eye swelling (Eye disorders) | 1/30 | 0/30
Eyelid oedema (Eye disorders) | 1/30 | 0/30
Vision blurred (Eye disorders) | 1/30 | 0/30
Diarrhoea (Gastrointestinal disorders) | 17/30 | 10/30
Abdominal pain (Gastrointestinal disorders) | 11/30 | 13/30
Nausea (Gastrointestinal disorders) | 11/30 | 10/30
Vomiting (Gastrointestinal disorders) | 14/30 | 7/30
Abdominal pain upper (Gastrointestinal disorders) | 5/30 | 8/30
Constipation (Gastrointestinal disorders) | 8/30 | 5/30
Stomatitis (Gastrointestinal disorders) | 7/30 | 6/30
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4/30 | 4/30
Flatulence (Gastrointestinal disorders) | 3/30 | 2/30
Abdominal distension (Gastrointestinal disorders) | 2/30 | 2/30
Abdominal discomfort (Gastrointestinal disorders) | 2/30 | 1/30
Abdominal pain lower (Gastrointestinal disorders) | 0/30 | 3/30
Dyspepsia (Gastrointestinal disorders) | 2/30 | 1/30
Oral pain (Gastrointestinal disorders) | 1/30 | 2/30
Dry mouth (Gastrointestinal disorders) | 1/30 | 1/30
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/30 | 1/30
Gingival bleeding (Gastrointestinal disorders) | 2/30 | 0/30
Gingival pain (Gastrointestinal disorders) | 1/30 | 1/30
Glossodynia (Gastrointestinal disorders) | 2/30 | 0/30
Rectal haemorrhage (Gastrointestinal disorders) | 0/30 | 2/30
Toothache (Gastrointestinal disorders) | 1/30 | 1/30
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1/30 | 0/30
Anal fissure (Gastrointestinal disorders) | 1/30 | 0/30
Anal pruritus (Gastrointestinal disorders) | 1/30 | 0/30
Ascites (Gastrointestinal disorders) | 1/30 | 0/30
Cheilitis (Gastrointestinal disorders) | 1/30 | 0/30
Dental caries (Gastrointestinal disorders) | 0/30 | 1/30
Dysphagia (Gastrointestinal disorders) | 0/30 | 1/30
Enterocutaneous fistula (Gastrointestinal disorders) | 0/30 | 1/30
Faeces discoloured (Gastrointestinal disorders) | 1/30 | 0/30
Food poisoning (Gastrointestinal disorders) | 1/30 | 0/30
Gastritis (Gastrointestinal disorders) | 1/30 | 0/30
Gastrointestinal perforation (Gastrointestinal disorders) | 1/30 | 0/30
Haemorrhoids (Gastrointestinal disorders) | 0/30 | 1/30
Intestinal obstruction (Gastrointestinal disorders) | 0/30 | 1/30
Lip swelling (Gastrointestinal disorders) | 0/30 | 1/30
Oesophagitis (Gastrointestinal disorders) | 0/30 | 1/30
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0/30 | 1/30
Peritonitis (Gastrointestinal disorders) | 1/30 | 0/30
Pneumatosis intestinalis (Gastrointestinal disorders) | 0/30 | 1/30
Stomach discomfort (Gastrointestinal disorders) | 1/30 | 0/30
Subileus (Gastrointestinal disorders) | 1/30 | 0/30
Tongue ulceration (Gastrointestinal disorders) | 1/30 | 0/30
Asthenia (General disorders) | 13/30 | 10/30
Fatigue (General disorders) | 12/30 | 10/30
Mucosal inflammation (General disorders) | 3/30 | 8/30
Oedema peripheral (General disorders) | 8/30 | 3/30
Pyrexia (General disorders) | 5/30 | 6/30
Chills (General disorders) | 3/30 | 4/30
Chest pain (General disorders) | 1/30 | 4/30
General physical health deterioration (General disorders) | 5/30 | 0/30
Disease progression (General disorders) | 1/30 | 3/30
Pain (General disorders) | 0/30 | 3/30
Death (General disorders) | 1/30 | 0/30
Face oedema (General disorders) | 1/30 | 0/30
Feeling hot (General disorders) | 0/30 | 1/30
Hernia pain (General disorders) | 1/30 | 0/30
Temperature intolerance (General disorders) | 1/30 | 0/30
Liver disorder (Hepatobiliary disorders) | 1/30 | 1/30
Hepatomegaly (Hepatobiliary disorders) | 0/30 | 1/30
Nasopharyngitis (Infections and infestations) | 3/30 | 1/30
Urinary tract infection (Infections and infestations) | 1/30 | 2/30
Herpes zoster (Infections and infestations) | 1/30 | 1/30
Wound infection (Infections and infestations) | 1/30 | 1/30
Bronchitis (Infections and infestations) | 0/30 | 1/30
Catheter related infection (Infections and infestations) | 0/30 | 1/30
Emphysematous cystitis (Infections and infestations) | 0/30 | 1/30
Folliculitis (Infections and infestations) | 1/30 | 0/30
Incision site cellulitis (Infections and infestations) | 1/30 | 0/30
Laryngitis (Infections and infestations) | 1/30 | 0/30
Pneumonia (Infections and infestations) | 1/30 | 0/30
Pyelonephritis (Infections and infestations) | 0/30 | 1/30
Sepsis (Infections and infestations) | 0/30 | 1/30
Septic shock (Infections and infestations) | 1/30 | 0/30
Tooth infection (Infections and infestations) | 1/30 | 0/30
Upper respiratory tract infection (Infections and infestations) | 0/30 | 1/30
Urinary tract infection staphylococcal (Infections and infestations) | 1/30 | 0/30
Vaginal infection (Infections and infestations) | 0/30 | 1/30
Contusion (Injury, poisoning and procedural complications) | 1/30 | 0/30
Fall (Injury, poisoning and procedural complications) | 1/30 | 0/30
Joint injury (Injury, poisoning and procedural complications) | 0/30 | 1/30
Muscle strain (Injury, poisoning and procedural complications) | 0/30 | 1/30
Blood thyroid stimulating hormone increased (Investigations) | 5/30 | 4/30
Weight decreased (Investigations) | 2/30 | 4/30
Blood alkaline phosphatase increased (Investigations) | 3/30 | 2/30
Aspartate aminotransferase increased (Investigations) | 2/30 | 2/30
Gamma-glutamyltransferase increased (Investigations) | 3/30 | 1/30
Alanine aminotransferase increased (Investigations) | 1/30 | 2/30
Blood creatinine increased (Investigations) | 2/30 | 0/30
Alanine aminotransferase (Investigations) | 0/30 | 1/30
Blood bilirubin increased (Investigations) | 0/30 | 1/30
Blood potassium decreased (Investigations) | 1/30 | 0/30
Blood urea increased (Investigations) | 1/30 | 0/30
Breath sounds absent (Investigations) | 0/30 | 1/30
Mean cell haemoglobin increased (Investigations) | 1/30 | 0/30
Mean cell volume abnormal (Investigations) | 1/30 | 0/30
Anorexia (Metabolism and nutrition disorders) | 8/30 | 7/30
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3/30 | 5/30
Hypokalaemia (Metabolism and nutrition disorders) | 2/30 | 2/30
Hypophosphataemia (Metabolism and nutrition disorders) | 2/30 | 1/30
Decreased appetite (Metabolism and nutrition disorders) | 2/30 | 0/30
Dehydration (Metabolism and nutrition disorders) | 1/30 | 1/30
Hyperkalaemia (Metabolism and nutrition disorders) | 1/30 | 1/30
Cachexia (Metabolism and nutrition disorders) | 1/30 | 0/30
Hyperglycaemia (Metabolism and nutrition disorders) | 0/30 | 1/30
Hypocalcaemia (Metabolism and nutrition disorders) | 1/30 | 0/30
Hyponatraemia (Metabolism and nutrition disorders) | 1/30 | 0/30
Back pain (Musculoskeletal and connective tissue disorders) | 7/30 | 6/30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9/30 | 2/30
Arthralgia (Musculoskeletal and connective tissue disorders) | 5/30 | 2/30
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4/30 | 3/30
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3/30 | 2/30
Myalgia (Musculoskeletal and connective tissue disorders) | 2/30 | 3/30
Bone pain (Musculoskeletal and connective tissue disorders) | 2/30 | 0/30
Flank pain (Musculoskeletal and connective tissue disorders) | 0/30 | 1/30
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1/30 | 0/30
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0/30 | 1/30
Neck pain (Musculoskeletal and connective tissue disorders) | 1/30 | 0/30
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1/30 | 0/30
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/30 | 0/30
Headache (Nervous system disorders) | 8/30 | 6/30
Dysgeusia (Nervous system disorders) | 3/30 | 2/30
Ageusia (Nervous system disorders) | 2/30 | 1/30
Dizziness (Nervous system disorders) | 2/30 | 1/30
Hyperaesthesia (Nervous system disorders) | 1/30 | 1/30
Hypogeusia (Nervous system disorders) | 2/30 | 0/30
Neuropathy peripheral (Nervous system disorders) | 2/30 | 0/30
Paraesthesia (Nervous system disorders) | 1/30 | 1/30
Amnesia (Nervous system disorders) | 0/30 | 1/30
Cerebrovascular accident (Nervous system disorders) | 0/30 | 1/30
Formication (Nervous system disorders) | 1/30 | 0/30
Psychomotor skills impaired (Nervous system disorders) | 1/30 | 0/30
Somnolence (Nervous system disorders) | 1/30 | 0/30
Syncope (Nervous system disorders) | 1/30 | 0/30
Transient ischaemic attack (Nervous system disorders) | 0/30 | 1/30
Tremor (Nervous system disorders) | 0/30 | 1/30
Depression (Psychiatric disorders) | 3/30 | 2/30
Insomnia (Psychiatric disorders) | 3/30 | 1/30
Anxiety (Psychiatric disorders) | 0/30 | 2/30
Confusional state (Psychiatric disorders) | 1/30 | 0/30
Dysuria (Renal and urinary disorders) | 1/30 | 2/30
Pollakiuria (Renal and urinary disorders) | 1/30 | 2/30
Renal impairment (Renal and urinary disorders) | 1/30 | 1/30
Renal pain (Renal and urinary disorders) | 2/30 | 0/30
Urinary tract disorder (Renal and urinary disorders) | 1/30 | 1/30
Haematuria (Renal and urinary disorders) | 1/30 | 0/30
Nephrotic syndrome (Renal and urinary disorders) | 0/30 | 1/30
Proteinuria (Renal and urinary disorders) | 0/30 | 1/30
Renal failure (Renal and urinary disorders) | 0/30 | 1/30
Urinary incontinence (Renal and urinary disorders) | 1/30 | 0/30
Breast pain (Reproductive system and breast disorders) | 1/30 | 1/30
Vaginal haemorrhage (Reproductive system and breast disorders) | 2/30 | 0/30
Menorrhagia (Reproductive system and breast disorders) | 1/30 | 0/30
Metrorrhagia (Reproductive system and breast disorders) | 1/30 | 0/30
Pelvic pain (Reproductive system and breast disorders) | 0/30 | 1/30
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1/30 | 0/30
Vulvovaginal dryness (Reproductive system and breast disorders) | 0/30 | 1/30
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7/30 | 5/30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3/30 | 4/30
Cough (Respiratory, thoracic and mediastinal disorders) | 0/30 | 5/30
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/30 | 2/30
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1/30 | 0/30
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0/30 | 1/30
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1/30 | 0/30
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0/30 | 1/30
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1/30 | 0/30
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/30 | 1/30
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1/30 | 0/30
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1/30 | 0/30
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8/30 | 7/30
Hair colour changes (Skin and subcutaneous tissue disorders) | 7/30 | 6/30
Rash (Skin and subcutaneous tissue disorders) | 6/30 | 2/30
Dry skin (Skin and subcutaneous tissue disorders) | 4/30 | 2/30
Eczema (Skin and subcutaneous tissue disorders) | 1/30 | 5/30
Yellow skin (Skin and subcutaneous tissue disorders) | 3/30 | 3/30
Pruritus (Skin and subcutaneous tissue disorders) | 4/30 | 0/30
Alopecia (Skin and subcutaneous tissue disorders) | 1/30 | 2/30
Skin discolouration (Skin and subcutaneous tissue disorders) | 1/30 | 2/30
Skin ulcer (Skin and subcutaneous tissue disorders) | 2/30 | 1/30
Dermatitis (Skin and subcutaneous tissue disorders) | 1/30 | 1/30
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/30 | 1/30
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0/30 | 2/30
Acne (Skin and subcutaneous tissue disorders) | 1/30 | 0/30
Blister (Skin and subcutaneous tissue disorders) | 1/30 | 0/30
Dermal cyst (Skin and subcutaneous tissue disorders) | 1/30 | 0/30
Erythema (Skin and subcutaneous tissue disorders) | 1/30 | 0/30
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1/30 | 0/30
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1/30 | 0/30
Nail disorder (Skin and subcutaneous tissue disorders) | 1/30 | 0/30
Rash macular (Skin and subcutaneous tissue disorders) | 1/30 | 0/30
Skin reaction (Skin and subcutaneous tissue disorders) | 0/30 | 1/30
Urticaria (Skin and subcutaneous tissue disorders) | 1/30 | 0/30
Sinus operation (Surgical and medical procedures) | 1/30 | 0/30
Hypertension (Vascular disorders) | 10/30 | 8/30
Capillary fragility (Vascular disorders) | 0/30 | 1/30
Hypertensive crisis (Vascular disorders) | 0/30 | 1/30
Pallor (Vascular disorders) | 0/30 | 1/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosure, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.